CLINICAL TRIAL: NCT03469180
Title: Comparison of Treadmill and Whole Body Vibration Training in Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Elif Durgut, Lecturer,MSc,PT, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvuedurgut01
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Treadmill Training; Whole Body Vibration Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Childrens in this group will receive treadmill training, three times a week for 8 weeks. Each season will be supervised and last 45 minutes.
  Interventions: Other: Treadmill training
- Training Group (Experimental): İn addition to treadmill training, childrens in this group (after a rest for 5 minutes) will also receive whole body vibration training for 15 minutes.
  Interventions: Other: Treadmill training; Other: Whole body vibration training

INTERVENTIONS:
Other: Treadmill training — Treadmill training Each season will be supervised and last 45 minutes. Treadmill speed will be adjusted to the child's maximal heart rate (MHR) (between 65 to 75 percent of the MHR).
Other: Whole body vibration training — Whole body vibration training whole body vibration frequence will be 50 Hertz and childrens will be standing position on vibration platform .
  Arms: Training Group

SUMMARY:
It is reported in the literature that children with attention deficit hyperactivity disorder (ADHD) may have executive function deficits, impaired social functions, emotional dysregulation, behavioral disorders and motor impairments. Furthermore, studies have shown that exercise, such as acute and chronic aerobic exercises and acute whole body vibration training, improves executive functions and motor abilities and so it is hypothesized that exercise may have a potential or additional treatment option for children with ADHD. Neurobiological researches have already proven the effects on brain changes during exercise and in the case of ADHD, increasing levels of serotonin, dopamine, and norepinephrine within the front striatal lobes of the brain were highlighted when discussing the effects on this neurodevelopmental disorder. The literature emphasizes the importance of physical activity in children with ADHD, but there is no clarity regarding the frequency, intensity or duration of the exercise. Thus, the aim of this study was to investigate and compare the effects of treadmill training as an aerobic exercise and whole body vibration training on executive functions and balance in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis (Previously not taking or not taking medication for ADHD)
* Being going to primary school

Exclusion Criteria:

* Having a chronic and serious medical condition

  * Seizure-like neurological impairment
  * Autism spectrum disorder, vision, speech, hearing problems

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-03-24 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline postural stability test score in Biodex Balance System at 8 weeks | Eight weeks
  The Postural Stability Training mode is designed to emphasize specific movement patterns or strategies by placing markers anywhere on the screen grid. The patient's score is a tally of how many times the patient can touch targets with the on-screen cursor during any session. Time counts up or down as set.The Postural Stability Test emphasizes a patient's ability to maintain center of balance. The patient's score on this test assesses deviations from center, thus a lower score is more desirable than a higher score.
Change from baseline limits of stability test score in Biodex Balance System at 8 weeks | Eight weeks
  The Limits of Stability Training screen is designed to challenge the user to move through a movement pattern consistent with the sway envelope.This test challenges patients to move and control their center of gravity within their base of support.
  During each test trial, patients must shift their weight to move the cursor from the center target to a blinking target and back as quickly and with as little deviation as possible. The same process is repeated for each of nine targets
Change from baseline sensory integration and balance test score in Biodex Balance System at 8 weeks | Eight weeks
Change from baseline single leg balance test score in Biodex Balance System at 8 weeks | Eight weeks
  The low stability level of four will challenge subjects and provide the data necessary to assess the subject's single leg postural stability

SECONDARY OUTCOMES:
Change from baseline Stroop test score at 8 weeks | Eight weeks
  This test assesses the response inhibition and measures the ability to shift perceptual set in accordance with changing demands. It also measures the inhibition of a habitual behavior pattern and behaving in an unusual manner. Defects in these abilities result in lack of perseveration, stereotypic behaviors, and difficulty in controlling behavior. These functions are mainly controlled by the frontal lobes. Higher interference scores indicate poorer performance. This test has been adapted and standardized for the Turkish population
Change from baseline BRIEF (Behavior Rating Inventory of Executive Function) score at 8 weeks | Eight weeks
  İt assesses executive function and self-regulation in children and teens. High scores indicate a higher level of dysfunction in a specific domain of executive functions.
Change from baseline Conners score at 8 weeks | Eight weeks
  The scale has been used for the identification of behaviour disorders in children. Higher scores describe more severe behaviour disorder
Change from baseline the Pediatric Quality of Life Inventory (PedsQL) score at 8 weeks | Eight weeks
  The Pediatric Quality of Life Inventory (PedsQL) is a modular instrument for measuring health related quality of life of 2-18 year-old-children. Higher scores indicate higher health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Elif Durgut, Msc,PT, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided